CLINICAL TRIAL: NCT01680991
Title: A Multi-Center, Open Label, Single Arm, Multiple Dose Study to Assess the Pharmacokinetics of RO5072759 in Chinese Patients With CD20+ Malignant Disease
Brief Title: A Study of Obinutuzumab in Chinese Participants With CD20+ Malignant Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YP25623
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-03

CONDITIONS: Lymphocytic Leukemia, Chronic, Diffuse Large B-cell Lymphoma, Follicular Lymphoma
MeSH Terms: conditions — Leukemia, Lymphoid; Bronchiolitis Obliterans Syndrome; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — obinutuzumab

ARMS (3):
- CLL: 1000 mg Obinutuzumab (Experimental): Participants with chronic lymphocytic leukemia (CLL) will receive 1000 milligrams (mg) obinutuzumab as an intravenous (IV) infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. The first infusion on Cycle 1 Day 1 will be given over two days: Day 1 and Day 2. Additional doses of obinutuzumab will be administered on Cycle 1 Day 8 and Day 15.
  Interventions: Drug: Obinutuzumab
- DLBCL: 1000 mg Obinutuzumab (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) will receive 1000 mg obinutuzumab as an IV infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab will be administered on Cycle 1 Day 8 and Day 15.
  Interventions: Drug: Obinutuzumab
- FL: 1000 mg Obinutuzumab (Experimental): Participants with follicular lymphoma (FL) will receive 1000 mg obinutuzumab as an IV infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab will be administered on Cycle 1 Day 8 and Day 15.
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — Multiple doses of obinutuzumab.
  Other Names: RO5072759; GA101

SUMMARY:
This multi-center, open-label, single-arm study will evaluate the pharmacokinetics and safety of obinutuzumab in participants with cluster of differentiation (CD) 20 positive (+) malignant disease. Participants will receive multiple doses of obinutuzumab. The anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20+ B-cell lymphoma or B-CLL
* Refractory/relapsed CLL, FL, and DLBCL
* At least 1 measurable lesion (greater than [>] 1.5 centimeters [cm] in its largest dimension) with the exception of CLL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy >6 months

Exclusion Criteria:

* Prior use of any investigational antibody therapy within 6 months of study start
* Prior use of any anti-cancer vaccine
* Prior administration of rituximab within 3 months of study start
* Prior administration of radioimmunotherapy 3 months prior to study entry
* Central nervous system lymphoma
* History of other malignancy
* Evidence of significant, uncontrolled concomitant disease
* Abnormal laboratory values
* Patients with progressive multifocalleukoencephalopathy (PML)
* Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- China (3):
  - Beijing
  - Guangzhou
  - Shanghai

REFERENCES:
- [Derived] Qin Y, Song Y, Shen Z, Du X, Ji W, Hsu W, Zhu J, Shi Y. Safety and efficacy of obinutuzumab in Chinese patients with B-cell lymphomas: a secondary analysis of the GERSHWIN trial. Cancer Commun (Lond). 2018 May 30;38(1):31. doi: 10.1186/s40880-018-0300-5. PMID 29843792
- [Derived] Zhai J, Qin Y, Zhu J, Song Y, Shen Z, Du X, Jamois C, Brewster M, Shi Y, Shi J. Pharmacokinetics of obinutuzumab in Chinese patients with B-cell lymphomas. Br J Clin Pharmacol. 2017 Jul;83(7):1446-1456. doi: 10.1111/bcp.13232. Epub 2017 Feb 14. PMID 28072473

RESULTS

PARTICIPANT FLOW:
Groups:
- CLL: 1000 mg Obinutuzumab: Participants with chronic lymphocytic leukemia (CLL) received 1000 milligrams (mg) obinutuzumab as an intravenous (IV) infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab were administered on Cycle 1 Day 8 and Day 15. The first infusion on Cycle 1 Day 1 was given over two days: Day 1- 100 mg and Day 2- 900 mg.
- DLBCL: 1000 mg Obinutuzumab: Participants with diffuse large B-cell lymphoma (DLBCL) received 1000 mg obinutuzumab as an IV infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab were administered on Cycle 1 Day 8 and Day 15.
- FL: 1000 mg Obinutuzumab: Participants with follicular lymphoma (FL) received 1000 mg obinutuzumab as an IV infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab were administered on Cycle 1 Day 8 and Day 15.
Period: Overall Study
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Started | 12 | 23 | 13
Completed | 4 | 4 | 9
Not Completed | 8 | 19 | 4
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Progressive disease (PD) | 0 | 10 | 0
Not completed — Physician Decision | 0 | 7 | 2
Not completed — Bad physical condition | 0 | 0 | 1
Not completed — PD confirmed in other hospital | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of study drug.
Groups:
- CLL: 1000 mg Obinutuzumab: Participants with CLL received 1000 mg obinutuzumab as an IV infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab were administered on Cycle 1 Day 8 and Day 15. The first infusion on Cycle 1 Day 1 was given over two days: Day 1- 100 mg and Day 2- 900 mg.
- DLBCL: 1000 mg Obinutuzumab: Participants with DLBCL received 1000 mg obinutuzumab as an IV infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab were administered on Cycle 1 Day 8 and Day 15.
- FL: 1000 mg Obinutuzumab: Participants with FL received 1000 mg obinutuzumab as an IV infusion, on Day 1 of each 21-day cycle for a maximum of 8 cycles. Additional doses of obinutuzumab were administered on Cycle 1 Day 8 and Day 15.
- Total: Total of all reporting groups
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab | Total
Number analyzed (Participants) | 12 | 23 | 13 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (12.0) | 53.3 (15.8) | 55.1 (8.8) | 55.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 5 | 22
  Male | 7 | 11 | 8 | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration Time Curve From Zero to Day 7 (AUC0-7) of Obinutuzumab on Day 1, Cycle 1
Description: DLBCL and FL are sub-types of Non-Hodgkin's Lymphoma (NHL) and time frame for these 2 groups was presented under NHL. For CLL, pharmacokinetic (PK) parameters were from Cycle 1 Day 1 and Day 2 dosing, due to split dosing.
Time Frame: Cycle 1-NHL: within 2 hours (h) pre-dose (Pr-D), end of infusion (EoI), 4, 24, 72 and 120 h post-infusion (Po-I) on Day 1; CLL: within 2 h Pr-D, EoI on Days 1,2; 4, 24, 72 and 120 h Po-I on Day 2. NHL and CLL: within 2 h Pr-D on Day 8
Population: PK analysis population included all participants who received at least 1 dose of study drug and had serum concentrations available. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*micrograms per milliliter
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 11 | 21 | 13
day*micrograms per milliliter | 1458 (34.8) | 1750 (20.5) | 1647 (20.7)

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Obinutuzumab on Day 1, Cycle 1
Description: DLBCL and FL are sub-types of NHL and time frame for these 2 groups was presented under NHL. For CLL, PK parameters were from Cycle 1 Day 1 and Day 2 dosing, due to split dosing.
Time Frame: Cycle 1-NHL: within 2 h Pr-D, EoI, 4, 24, 72 and 120 h Po-I on Day 1; CLL: within 2 h Pr-D, EoI on Days 1,2; 4, 24, 72 and 120 h Po-I on Day 2. NHL and CLL: within 2 h Pr-D on Day 8
Population: PK analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 11 | 21 | 13
micrograms per milliliter (mcg/mL) | 369 (31.8) | 442 (21.1) | 437 (16.7)

3. Primary Outcome: Area Under the Serum Concentration Versus Time Curve From 0 to Day 21 (AUC0-21) of Obinutuzumab at Cycle 8
Time Frame: Cycle 8: within 2 h Pr-D, EoI, 4, 24, 72, 120, 168, 336 (Day 15), and 504 (Day 22) h Po-I on Day 1
Population: PK analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 9 | 8 | 11
day*mcg/mL | 12289 (42.7) | 13000 (37.3) | 11285 (26.7)

4. Primary Outcome: Cmax of Obinutuzumab at Cycle 8
Time Frame: Cycle 8: within 2 h Pr-D, EoI, 4, 24, 72, 120, 168, 336 (Day 15), and 504 (Day 22) h Po-I on Day 1
Population: PK analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 9 | 8 | 11
mcg/mL | 1050 (32.6) | 966 (28.3) | 867 (19.6)

5. Secondary Outcome: Time to Maximum Observed Serum Concentration (Tmax) of Obinutuzumab at Cycle 8
Time Frame: Cycle 8: within 2 h Pr-D, EoI, 4, 24, 72, 120, 168, 336 (Day 15), and 504 (Day 22) h Po-I on Day 1
Population: PK analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 9 | 8 | 11
hours | 3.5 [3.3 to 25.5] | 7.25 [3.3 to 27.5] | 4.0 [3.2 to 7.8]

6. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Description: Half-life is the time measured for the serum concentration of study drug to decrease (Dec) by one half.
Time Frame: Cycle 8: within 2 h Pr-D, EoI, 4, 24, 72, 120, 168, 336 (Day 15), and 504 (Day 22) h Po-I on Day 1, 4-week follow-up (Day 29), 3 and 6 months after Cycle 8 dosing
Population: PK analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 9 | 6 | 11
day | 21.5 (71.8) | 33.3 (68.6) | 26.7 (49.6)

7. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Obinutuzumab at Cycle 8
Description: Vss reflects the actual blood and tissue volume into which a drug is distributed and the relative binding of drug to protein in these spaces.
Time Frame: Cycle 8: within 2 h Pr-D, EoI, 4, 24, 72, 120, 168, 336 (Day 15), and 504 (Day 22) h Po-I on Day 1
Population: PK analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 9 | 6 | 11
Liter | 3.32 (27.9) | 4.49 (38.2) | 4.03 (21.5)

8. Secondary Outcome: Total Systemic Clearance at Steady State (CLss) of Obinutuzumab at Cycle 8
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Cycle 8: within 2 h Pr-D, EoI, 4, 24, 72, 120, 168, 336 (Day 15), and 504 (Day 22) h Po-I on Day 1
Population: PK analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 9 | 8 | 11
mL/day | 81.4 (42.7) | 76.9 (37.3) | 88.6 (26.7)

9. Secondary Outcome: Minimum Observed Serum Concentration of Obinutuzumab
Time Frame: Within 2 hours Pr-D on Day 1 of Cycles 2-8 and on Days 8,15 of Cycle 1
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome and "n" is the number of participants evaluable at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 11 | 22 | 13
mcg/mL
  Cycle 1-Day 8 (n=11,22,13) | 156 (57.2) | 186 (25.2) | 148 (39.2)
  Cycle 1-Day 15 (n=11,22,13) | 282 (69.4) | 350 (23.7) | 284 (26.5)
  Cycle 2 (n=11,21,13) | 389 (71.2) | 458 (26.3) | 433 (31.2)
  Cycle 3 (n=10,18,13) | 260 (246) | 367 (49.6) | 346 (31)
  Cycle 4 (n=10,14,13) | 232 (279.7) | 370 (49.2) | 346 (31)
  Cycle 5 (n=9,11,11) | 299 (91.2) | 412 (42) | 396 (44.8)
  Cycle 6 (n=9,10,11) | 317 (93.5) | 425 (38.2) | 361 (40.6)
  Cycle 7 (n=9,10,11) | 358 (80.6) | 367 (40.3) | 375 (41.3)
  Cycle 8 (n=9,8,11) | 403 (85.3) | 455 (45.4) | 352 (38.4)

10. Secondary Outcome: Percentage of Participants With Complete Response (CR), CR Unconfirmed (CRu) at End of Treatment (1 Month After Cycle 8) in NHL Participants (DLBCL and FL Participants) Per Cheson 1999 Criteria
Description: CR: 1) Disappearance of clinical and radiographic evidence of disease, related symptoms and normalization of biochemical abnormalities definitely assignable to NHL, 2) Lymph nodes (LN) and nodal masses regressed to normal size after therapy (AT) (≤1.5 centimeters [cm] in their greatest transverse diameter [GTD] for LN greater than (>) 1.5 cm before therapy [BT]). LN that were 1.1 to 1.5 cm in their GTD BT decreased to ≤1 cm in GTD AT, or >75% in the sum of the products (SPD) of the GTD, 3) Enlarged spleen regressed in size and not palpable, 4) Absence of macroscopic nodules, 5) Enlarged organs decreased in size, and 6) If the bone marrow (BM) was involved, the infiltrate must be cleared on repeat BM aspirate and biopsy. CRu included those participants who met CR Criteria 1 and 3, but with 1 or more of the following features: a) A residual LN mass >1.5 cm in GTD that has regressed by more than 75% in their SPD, and b) Indeterminate BM (increased [Inc] number or size of aggregates).
Time Frame: 1 month after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for DLBCL and FL arm groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 23 | 13
percentage of participants
  CR | 0 [0.00 to 14.82] | 0 [0.00 to 24.71]
  CRu | 4.3 [0.11 to 21.95] | 0 [0.00 to 24.71]

11. Secondary Outcome: Percentage of Participants With Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD) at End of Treatment (1 Month After Cycle 8) in NHL Participants (DLBCL and FL Participants) Per Cheson 1999 Criteria
Description: PR: 1) ≥50% decrease in SPD of the 6 largest dominant nodes/nodal masses. These nodes or masses selected according to the following features: a) clearly measurable in ≥2 perpendicular dimensions, b) from as disparate regions of the body as possible, and c) included mediastinal and retroperitoneal areas of disease. 2) No increase in size of other nodes (liver/spleen). 3) Splenic and hepatic nodules regressed by ≥50% in SPD. 4) With exception of splenic and hepatic nodules, involvement of other organs was considered assessable and not measurable disease. 5) BM assessment is irrelevant for determination of a PR because it was assessable and not measurable disease; however, if positive, the cell type was specified. 6) No new sites of disease. PD requires the following: 1) ≥50% increase from nadir in the SPD of any previously identified abnormal node for PRs or nonresponders. 2) Appearance of any new lesion during or at the end of therapy. SD is defined as less than a PR but not PD.
Time Frame: 1 month after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for DLBCL and FL arm groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 23 | 13
percentage of participants
  PR | 8.7 [1.07 to 28.04] | 46.2 [19.22 to 74.87]
  SD | 8.7 [1.07 to 28.04] | 30.8 [9.09 to 61.43]
  PD | 65.2 [42.73 to 83.62] | 23.1 [5.04 to 53.81]

12. Secondary Outcome: Percentage of Participants With Best Overall Response (BOR) of CR, CRu at Anytime During Study in NHL Participants (DLBCL and FL Participants) Per Cheson 1999 Criteria
Description: CR: 1) Disappearance of clinical and radiographic evidence of disease, related symptoms and normalization of biochemical abnormalities definitely assignable to NHL, 2) LN and nodal masses regressed to normal size AT (≤1.5 cm] in their GTD for LN >1.5 cm BT). LN that were 1.1 to 1.5 cm in their GTD BT decreased to ≤1 cm in GTD AT, or >75% in the SPD of the GTD, 3) Enlarged spleen regressed in size and not palpable, 4) Absence of macroscopic nodules in any organs, 5) Enlarged organs decreased in size, and 6) If the BM was involved, the infiltrate must be cleared on repeat BM aspirate and biopsy. CRu included those participants who met CR Criteria 1 and 3, but with 1 or more of the following features: a) A residual LN mass >1.5 cm in GTD that has regressed by more than 75% in their SPD, b) Indeterminate BM (increased number or size of aggregates).
Time Frame: From screening to up to 1 month after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for DLBCL and FL arm groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 23 | 13
percentage of participants
  CR | 0 [0.00 to 14.82] | 0 [0.00 to 24.71]
  CRu | 4.3 [0.11 to 21.95] | 0 [0.00 to 24.71]

13. Secondary Outcome: Percentage of Participants With BOR of PR, SD, and PD at Anytime During Study in NHL Participants (DLBCL and FL Participants) Per Cheson 1999 Criteria
Description: as for outcome 11
Time Frame: From screening to up to 1 month after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for DLBCL and FL arm groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 23 | 13
percentage of participants
  PR | 21.7 [7.46 to 43.70] | 61.5 [31.58 to 86.14]
  SD | 26.1 [10.23 to 48.41] | 30.8 [9.09 to 61.43]
  PD | 39.1 [19.71 to 61.46] | 7.7 [0.19 to 36.03]

14. Secondary Outcome: Percentage of Participants With Complete Remission (CRe), CRe With Incomplete BM Recovery (CRi) at End of Treatment (1 Month After Cycle 8) in CLL Participants According to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Guidelines
Description: CRe required the following criteria as assessed, at least 2 months from completing therapy: a) peripheral blood lymphocytes (PBL) less than (<) 4 x 10^9/L, b) Absence of significant lymphadenopathy (LD) by physical examination (PE), c) No hepatomegaly/splenomegaly (HM/SM) by PE, d) Absence of constitutional symptoms and e) Blood counts above the following values (i. Neutrophils [Neu] >1.5 x 10^9/L without the need for exogenous growth factors [EGF], ii. Platelets (Plt) >100 x 10^9/L without the need for EGF, and iii. Hemoglobin (Hb) >11.0 g/dL without blood transfusion or need for erythropoietin), and d) Once clinical and laboratory reports demonstrated CRe, a BM aspirate and biopsy was performed at least 2 months after the last treatment; to define a CRe, BM sample should be normocellular for age, <30% of the cells being PBL and lymphoid nodules absent. CRi: CRe but persistent anemia/thrombocytopenia/neutropenia unrelated to CLL, but related to drug toxicity.
Time Frame: 2 months after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for CLL participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 12
percentage of participants
  CRe | 0 [0.00 to 26.46]
  CRi | 0 [0.00 to 26.46]

15. Secondary Outcome: Percentage of Participants With PR, SD, and PD at End of Treatment (1 Month After Cycle 8) in CLL Participants According to IWCLL 2008 Guidelines
Description: Group A: a)Dec LN size by ≥50% either in SPD of 6 LN or largest diameter of enlarged LN (ELN) detected BT, b)Reduction (Red) in BT enlargement of liver, c)Red in BT enlargement of spleen, d)Dec in PBL by ≥50% from baseline, e)A 50% Red in BM infiltrate or B-lymphoid nodules in BM and f)No Inc in any LN and no new ELN. Group B: a)Plt count=100,000/µL or Inc of ≥50% over baseline, b)Hb >11 g/dL or ≥50% Inc over baseline, c)Neu > 1500/µL or > 50% Inc over baseline. PR is considered as achieved if 2 of Group A criteria and 1 of Group B criteria were met for ≥2 months. PD is defined as LD (appearance of new lesion [ELN], SM, HM or other organ infiltrates) or Inc by ≥50% in greatest determined diameter of any previous site or Inc in previously noted enlargement of liver/spleen by ≥50% or new appearance of HM/SM or an Inc in number of PBL ≥50% or transformation to a more aggressive histology or occurrence of cytopenia attributable to CLL. SD is defined as less than a PR but is not PD.
Time Frame: 2 months after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for CLL participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 12
percentage of participants
  PR | 58.3 [27.67 to 84.83]
  SD | 8.3 [0.21 to 38.48]
  PD | 16.7 [2.09 to 48.41]

16. Secondary Outcome: Percentage of Participants With BOR of CRe, CRi at Anytime During the Study in CLL Participants According to IWCLL 2008 Guidelines
Description: CRe required the following criteria as assessed, at least 2 months from completing therapy: a) PBL <4 x 10^9/L, b) Absence of significant LD by PE, c) No HM/SM by PE, d) Absence of constitutional symptoms and e) Blood counts above the following values (i. Neu >1.5 x 10^9/L without the need for EGF, ii. Plt >100 x 10^9/L without the need for EGF, and iii. Hb >11.0 g/dL without blood transfusion or need for EGF, and d) Once clinical and laboratory reports demonstrated CRe, a BM aspirate and biopsy was performed at least 2 months after the last treatment; to define a CRe, BM sample should be normocellular for age, <30% of the cells being PBL and lymphoid nodules absent. CRi: CRe but persistent anemia/thrombocytopenia/neutropenia unrelated to CLL, but related to drug toxicity.
Time Frame: From screening to up to 2 months after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for CLL participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 12
percentage of participants
  CRe | 0 [0.00 to 26.46]
  CRi | 0 [0.00 to 26.46]

17. Secondary Outcome: Percentage of Participants With BOR of PR, SD, and PD at Anytime During Study in CLL Participants According to IWCLL 2008 Guidelines
Description: Group A: a)Dec LN size by ≥50% either in SPD of 6 LN or largest diameter of ELN detected BT, b)Red in BT enlargement of liver, c)Red in BT enlargement of spleen, d)Dec in PBL by ≥50% from baseline, e)A 50% Red in BM infiltrate or B-lymphoid nodules in BM and f)No Inc in any LN and no new ELN. Group B: a)Plt count=100,000/µL or Inc of ≥50% over baseline, b)Hb >11 g/dL or ≥50% Inc over baseline, c)Neu > 1500/µL or > 50% Inc over baseline. PR is considered as achieved if 2 of Group A criteria and 1 of Group B criteria were met for ≥2 months. PD is defined as LD (appearance of new lesion [ELN], SM, HM or other organ infiltrates) or Inc by ≥50% in greatest determined diameter of any previous site or Inc in previously noted enlargement of liver/spleen by ≥50% or new appearance of HM/SM or an Inc in number of PBL ≥50% or transformation to a more aggressive histology or occurrence of cytopenia attributable to CLL. SD is defined as less than a PR but is not PD.
Time Frame: From screening to up to 2 months after the last dose (received on Day 148) of study drug
Population: Safety analysis population. Data reported only for CLL participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 12
percentage of participants
  PR | 75.0 [42.81 to 94.51]
  SD | 8.3 [0.21 to 38.48]
  PD | 0 [0.00 to 26.46]

18. Secondary Outcome: Number of Participants With Positive Human Anti-Human Antibodies (HAHA)
Description: For the detection of HAHA, serum samples were initially analyzed using a validated enzyme linked immunosorbent assay (ELISA) method (screening assay, tier 1). The lower limit of quantification (LLOQ) in undiluted serum was 18.4 nanograms per milliliter (ng/mL). The precision ranged from 4.85 percent (%) to 16.0%. In serum samples found positive, the presence of specific anti-obinutuzumab antibodies was confirmed or excluded using the same ELISA method with an appropriate immunocompetition step (addition of excess obinutuzumab, confirmation assay, tier 2). Samples were confirmed as containing specific anti-obinutuzumab antibodies if there was a signal reduction ≥85.7% in the presence of obinutuzumab.
Time Frame: Cycle 1 (Day 1), Cycle 4 (Day 1), 4-week follow-up, 3 and 6 month follow-up
Population: Safety analysis population. "n" represents the number of participants who were evaluable at the specified time point.
Measure: Number; unit: participants
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 12 | 23 | 13
participants
  Cycle 1, Day 1 (n=12,23,13) | 0 | 0 | 0
  Cycle 4, Day 1 (n=11,14,13) | 0 | 0 | 0
  4 week follow-up (n=10,10,11) | 0 | 0 | 0
  3 month follow-up (n=8,4,11) | 0 | 0 | 0
  6 month follow-up (n=7,4,11) | 0 | 0 | 1

19. Secondary Outcome: Number of Participants With Positive Human Anti-Chimeric Antibodies (HACA)
Description: Serum concentrations of HACA against rituximab were determined by ELISA. The LLOQ in undiluted serum was 5.00 relative units per milliliter (RU/mL). The precision and accuracy of the assay, as determined from the analysis of quality control samples, were satisfactory throughout the study; precision ranged from 6.4% to 13.6% and accuracy ranged from 88.2% to 94.8%.
Time Frame: Cycle 1, Day 1
Population: Safety analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 10 | 20 | 7
participants | 2 | 1 | 0

20. Secondary Outcome: Number of Participants With B-cell Depletion or Recovery
Description: Depletion is defined as cluster of differentiation (CD) 19+ B-cell count <0.07 x10^9/L.Recovery is defined as CD19+ B-cell equal to or greater than 0.07 x 10^9/L.
Time Frame: Screening, Cycle 1 (Days 1,8), Cycle 2 (Day 1), Cycle 4 (Day 1), Cycle 6 (Day 1), Cycle 8 (Day 1), 4 weeks after last dose of study drug and every 3 months after last dose of study drug up to 1 year
Population: Safety analysis population.
Measure: Number; unit: participants
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 12 | 23 | 13
participants
  B-cell Depletion | 9 | 23 | 13
  B-cell Recovery | 4 | 1 | 1

21. Secondary Outcome: Duration of Depletion of CD19+ B-cell
Description: Depletion is defined as CD19+ B-cell count < 0.07 x 10^9/L. The duration of depletion is defined as the number of days between first assessment of B-cell depletion and the first assessment where CD19+ cell count returned to at least the depletion level from baseline and not followed by any further B-cell depletion. If participant did not return to above depletion level, then the cut off is at the time of last assessment.
Time Frame: as for outcome 20
Population: Safety analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 9 | 23 | 12
days | 238.7 (182.5) | 141.0 (167.5) | 386.0 (176.0)

22. Secondary Outcome: Time to Recovery of CD19+ B-cell
Description: Recovery is defined as CD19+ B-cell equal to or greater than 0.07 x 10^9/L. Time to recovery is defined as time between the beginning of depletion and first value after end of treatment that is equal or above 0.07x10^9/L and not exclusively followed by depleted values only. If participant did not return to above recovery level then set to Null.
Time Frame: as for outcome 20
Population: Safety analysis population. Here, number of participants analyzed = participants who were evaluable for this outcome and "n" represents the number of participants evaluable for the specified category.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Number analyzed (Participants) | 4 | 1 | 1
days
  Time to recovery with PD (n=1,0,1) | 419 (NA) — Standard deviation is not applicable as data of a single participant is reported. | NA (NA) — No participant experienced B-cell recovery for this category. | 331.0 (NA) — Standard deviation is not applicable as data of a single participant is reported.
  Time to recovery without PD (n=3,1,0) | 229.0 (87.5) | 515.0 (NA) — Standard deviation is not applicable as data of a single participant is reported. | NA (NA) — No participant experienced B-cell recovery for this category.

ADVERSE EVENTS:
Time Frame: Until 3 months after last study drug (Up to approximately 9 months)
Description: Safety analysis population.
Arm/Group | CLL: 1000 mg Obinutuzumab | DLBCL: 1000 mg Obinutuzumab | FL: 1000 mg Obinutuzumab
Serious Adverse Events (participants affected / at risk) | 5/12 | 3/23 | 1/13
Other Adverse Events (participants affected / at risk) | 10/12 | 17/23 | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLL: 1000 mg Obinutuzumab (N=12) | DLBCL: 1000 mg Obinutuzumab (N=23) | FL: 1000 mg Obinutuzumab (N=13)
Pneumonia (Infections and infestations) | 2 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Submandibular mass (General disorders) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLL: 1000 mg Obinutuzumab (N=12) | DLBCL: 1000 mg Obinutuzumab (N=23) | FL: 1000 mg Obinutuzumab (N=13)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 | 5 | 3
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pyrexia (General disorders) | 6 | 3 | 2
Chills (General disorders) | 3 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Epididymitis (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Scleral haemorrhage (Eye disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.